CLINICAL TRIAL: NCT01454778
Title: Effects of Paclitaxel on Intimal Hyperplasia Status Post Lower Extremity Revascularization
Brief Title: Effects of Paclitaxel on Intimal Hyperplasia
Acronym: Pac1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Patrick Kelly (Other)
Responsible Party: Sponsor-Investigator, Patrick Kelly, Principal Investigator, Sanford Health
Organization: Sanford Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pac 1
Record Dates: First submitted 2011-04-04; First posted 2011-10-19 (Estimated); Results first posted 2016-05-24 (Estimated); Last update posted 2016-05-24 (Estimated); Status verified 2016-04

CONDITIONS: Peripheral Vascular Disease
Keywords: restenosis; peripheral vascular disease; lower extremity ischemia; claudication
MeSH Terms: conditions — Peripheral Vascular Diseases; Intermittent Claudication | interventions — Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel (Experimental)
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Paclitaxel — Paclitaxel in addition to angioplasty, stenting or atherectomy Dosing will be based on the lesion surface area, and will be calculated using the following formula: dose= 22/7 X diameter (mm) X length (mm) X 3 micrograms/mm^3
  Paclitaxel Dosage:
  Superficial Femoral/Common Femoral: 2.4 mg/inflation of balloon* Popliteal: 1.8 mg/inflation of balloon* Tibial: 1.4 mg/inflation of balloon*
  * not to exceed 10mg total dose
  Other Names: Taxol, Onxol

SUMMARY:
This is a single, one time, limited dose infusion of Paclitaxel, that will potentially prevent recurrent stenosis secondary to intimal hyperplasia when compared to the control group at 10 months.

DETAILED DESCRIPTION:
The investigators study consists of enrolling subjects that are already scheduled to have the blood vessels in their legs re-opened. The entire study is considered standard of care, except the administration of Paclitaxel. Subjects will be consented prior to any study related procedures and prior to procedure. Subjects that meet inclusion/exclusion and the infusion of Paclitaxel has been given, will then be enrolled in the study. After the plaque area has been treated with either angioplasty (inflation of a balloon compacting it against the artery wall), stent (a wire mesh tube that presses the plaque against the artery wall and opens the artery), and/or atherectomy(removal of plaque from the artery), Dr Kelly, Dr. Schultz, Dr, Laurich, or Dr. Santos will then use an infusion balloon (a balloon with an outer layer that has holes that allows a medication to be given) to administer the Paclitaxel. Every time the infusion balloon is blown up, a single dose of medication (Paclitaxel) will be applied to the target lesion. This will be repeated until all of the target lesions have been treated or a maximum dose of 10 mg of Paclitaxel has been given. All persons enrolled in this study will be treated with Paclitaxel. Subjects are expected to attend all follow up visits. These visits would occur even if the subject were not on the trial. Ankle-brachial index (ABI) (done by measuring blood pressure at the ankle and in the arm while a person is at rest. This test indicates if leg blockages are present) and Duplexes (An ultrasound that measures blood flow rates through the vessels. This test will indicate if leg blockages are present) will be done at the follow up visits. Both of these tests and all follow up visits are considered standard of care and will be charged to the subject or subject's insurance.

ELIGIBILITY:
Inclusion Criteria:

* ability to provide informed consent
* age 18-90 years old
* Rutherford 1-6
* occlusion or stenosis in the infrainguinal vessels

Exclusion Criteria:

* inability to pass the guide wire across the lesion
* pregnant or lactating women
* specific limb has not been previously treated with endovascular intervention

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-04; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Kelly, MD, Principal Investigator — Sanford Vascular Associates
Locations (1):
- Sanford Vascular Associates, Sioux Falls, South Dakota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Paclitaxel
Started | 50
Completed | 47
Not Completed | 3
Not completed — Lost to Follow-up | 2
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
Age, Customized [Mean (Full Range); unit: years] | 71.5 [44 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 35
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Stenosis Lower Extremity Post Revascularization Using Ankle-Brachial Index Measurement at 10 Months
Description: The Ankle-Brachial Index is calculated as a ratio of the ankle blood pressure and the arm blood pressure. The ABI and Rutherford Classification will be assessed at 10 months post revascularization
Time Frame: 10 months
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Paclitaxel: Paclitaxel: Paclitaxel coating in addition to angioplasty, stenting or atherectomy Dosing will be based on the lesion surface area, and will be calculated using the following formula: dose= 22/7 X diameter (mm) X length (mm) X 3 micrograms/mm^3
  Paclitaxel Dosage:
  Superficial Femoral/Common Femoral: 2.4 mg/inflation of balloon* Popliteal: 1.8 mg/inflation of balloon* Tibial: 1.4 mg/inflation of balloon*
  * not to exceed 10mg total dose
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
ratio | 0.93 (0.22)

2. Secondary Outcome: Freedom From Amputation Event
Time Frame: up to 10 months
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
percentage of participants | 100

3. Secondary Outcome: Freedom From Target Vessel Revascularization Event
Time Frame: up to 10 months
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
percentage of participants | 86

4. Secondary Outcome: Freedom From Binary Restenosis
Time Frame: 10 months
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
percentage of participants | 80

5. Secondary Outcome: Number of Serious Adverse Events
Time Frame: Up to 19 months
Measure: Number; unit: Number of SAE's
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
Number of SAE's | 2

6. Primary Outcome: Rutherford Classification of Peripheral Arterial Disease
Description: Evidence of stenosis of lower extremity as measured by the Rutherford Classification post revascularization. The ABI and Rutherford Classification will be assessed at 10 months post revascularization with a lower Rutherford score indicating a better outcome.
  0 = Asymptomatic, 1 = Mild Claudication, 2 = Moderate Claudication, 3 = Severe Claudication, 4 = Ischemic Rest Pain, 5 = Minor Tissue Loss, 6 = Ulceration or Gangrene
Time Frame: 10 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paclitaxel
Number analyzed (Participants) | 50
units on a scale | 0.63 (0.95)

ADVERSE EVENTS:
Arm/Group | Paclitaxel
Serious Adverse Events (participants affected / at risk) | 2/50
Other Adverse Events (participants affected / at risk) | 37/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=50)
Toe embolism (Vascular disorders) | 1 (1)
Restenosis of target lesion (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel (N=50)
Psuedoaneurysm (Vascular disorders) | 3 (3)
DVT (Vascular disorders) | 1 (1)
Occlusion (Vascular disorders) | 3 (3)
Dissection (Vascular disorders) | 8 (8)
Re-stenosis in the treated limb (Vascular disorders) | 16 (16)
Poor wound healing (Vascular disorders) | 2 (2)
Pain (Injury, poisoning and procedural complications) | 1 (1)
Claudication (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes